CLINICAL TRIAL: NCT00150072
Title: Phase II Study of Imatinib Mesylate in Chordoma
Brief Title: Efficacy and Safety of Imatinib in Chordoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BIT15
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chordoma
Keywords: chordoma; imatinib; PDGFR
MeSH Terms: conditions — Chordoma | interventions — Imatinib Mesylate

ARMS (1):
- imatinib (Experimental)
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: imatinib

SUMMARY:
Preliminary response data, observed by Casali (Cancer, 2004) with imatinib 800 mg/day in patients affected by chordoma, need to be confirmed by a Phase II study, whose primary endpoint will be the formal assessment of clinical and pathological response. Aim of the study will be to explore treatment's activity, but also the potential impact of tumor response, the feasibility and outcome of subsequent surgery and radiotherapy. In addition, patterns of tumour response need to be investigated as well, given the peculiar patterns of response shown with molecular-targeted therapy in solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of chordoma.
2. Biomolecular or immunohistochemical evidence of Imatinib mesylate target (PDGFRβ activation and/or presence of PDGFB). Biomolecular assessment of PDGFRβ activation should be made whenever possible. To this end, if frozen material is not available, obtaining of, fresh material is encouraged, if it should be obtained with no major distress for the patient, preferably through an incisional biopsy (to allow immunoprecipitation) or, if this is not feasible, a Trucut biopsy (to allow Western Blot assessment). However, if frozen or fresh material cannot be obtained, paraffined material is also acceptable.

   The biomolecular assessment will be centralized to the reference centers (to be defined).
3. Measurable or evaluable disease
4. Surgical resection of local disease unfeasible radically, or unaccepted by the patient, or amenable to become less demolitive, or easier, or likely more feasible, after cytoreduction, and/or metastatic disease. Debulking surgery before enrolment is allowed. In this case, enrolment should occur at least one month after surgery
5. Performance status 0, 1, 2 or 3 (ECOG) (see § 8.1).
6. Adequate end organ function, defined as the following: total bilirubin <1.5 x ULN, SGOT and SGPT <2.5 x UNL (or <5 x ULN if hepatic metastases are present), creatinine <1.5 x ULN.
7. Adequate bone marrow function, defined as the following: ANC >1.5 x 10^9/L, platelets >100 x 10^9/L, Hb >9 g/dL. Blood transfusions are allowed to reach the baseline requested Hb level.
8. Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
9. Written, voluntary, informed consent.

Exclusion Criteria:

1. Previous treatment with any other investigational or not investigational agents within 28 days of first day of study drug dosing.
2. Other primary malignancy with <5 years clinically assessed disease-free interval, except basal cell skin cancer, cervical carcinoma in situ, or other neoplasms judged to entail a low risk of relapse.
3. Grade III/IV cardiac problems as defined by the New York Heart Association Criteria (i.e., congestive heart failure, myocardial infarction within 6 months of study)
4. Severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
5. Known brain metastasis.
6. Known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
7. Known diagnosis of human immunodeficiency virus (HIV) infection.
8. Previous radiotherapy to >=25 % of the bone marrow.
9. Major surgery within 2 weeks prior to study entry.
10. Expected non-compliance to medical regimens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Tumor response | Every 3 months for 2 years
  objective response according to RECIST and clinical response

SECONDARY OUTCOMES:
Overall survival | 2 years
  from the first day of sudy treatment to the day of death for any cause
Progression free survival | 2 years
  from the first day of sudy treatment to the day of death for any cause or documented progression
Safety and tolerability | 2 years
  frequency of adverse events, abnormal lab values, bone pain, use of analgesic medication
proportion of patients undergoing complete surgery | 2 years
  number of pts undergoing complete surgery vs the one of pts not amenable to complete surgery at enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Italy (11):
  - Novartis Investigative Site, Aviano
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Candiolo
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Rozzano
  - Novartis Investigative Site, Torino
- Novartis Investigative Site, Lausanne, Switzerland

REFERENCES:
- [Result] Koren-Michowitz M, le Coutre P, Duyster J, Scheid C, Panayiotidis P, Prejzner W, Rowe JM, Schwarz M, Goldschmidt N, Nagler A. Activity and tolerability of nilotinib: a retrospective multicenter analysis of chronic myeloid leukemia patients who are imatinib resistant or intolerant. Cancer. 2010 Oct 1;116(19):4564-72. doi: 10.1002/cncr.25351. PMID 20572041